CLINICAL TRIAL: NCT03225989
Title: Phase I/II Trial Investigating an Immunostimulatory Oncolytic Adenovirus for Cancer
Brief Title: Trial Investigating an Immunostimulatory Oncolytic Adenovirus for Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lokon Pharma AB (Industry)
Collaborators: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LOKON002
Record Dates: First submitted 2017-07-04; First posted 2017-07-21 (Actual); Results first posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-10

CONDITIONS: Pancreatic Adenocarcinoma; Ovarian Cancer; Biliary Carcinoma; Colorectal Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants treated with LOAd703 at three dose levels (5x10e10 VP, 1x10e11 VP, 5x10e11 VP) and SOC tailored to the indication
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- LOAd703 (Experimental): LOAd703 oncolytic adenovirus administered add-on to standard of care chemotherapy or gemcitabine immune-conditioning if standard of care is no longer an option (e.g. after last line)
  Interventions: Drug: LOAd703

INTERVENTIONS:
Drug: LOAd703 — Oncolytic adenovirus serotype 5/35 encoding TMZ-CD40L and 4-1BBL

SUMMARY:
This Phase I/II trial evaluates LOAd703 in patients with cancer (pancreatic, biliary, colorectal or ovarian) together with their standard of care chemotherapy or using gemcitabine immune-conditioning. LOAd703 is administered by intratumoral image-guided injections. Maximum 50 patients can be enrolled.

LOAd703 is an immunostimulatory gene therapy using an selection replication competent adenovirus as a gene vehicle. The virus is derived from serotype 5 adenovirus with the fiber from serotype 35. It expresses the transgenes trimerized membrane-bound isoleucine zipper (TMZ) TMZ-CD40L and 41BBL under control of a cytomegalovirus (CMV) promoter.

DETAILED DESCRIPTION:
The trial is a Phase I/II trial evaluating the effect of LOAd703 in patients with pancreatic cancer, biliary cancer, ovarian cancer and colorectal cancer. LOAd703 is an oncolytic adenovirus serotype 5/35 encoding immunostimulatory transgenes: TMZ-CD40L and 41BBL. In Phase I, three doses (total viral load - 1x10e11, 5x10e11, 1x10e12 viral particles (VP)) of LOAd703 will be tested as add-on to standard of care or immune-conditioning gemcitabine chemotherapy. 8 treatments of LOAd703 will be delivered by image-guided intratumoral injection at the same time of chemotherapy. In Phase II stage of the study, patients will be treated at maximum tolerated dose/maximum tolerated study dose as defined in the Phase I stage. In both phases: tumor biopsies, blood samples and radiological imaging will be performed to evaluate safety, effect and mechanisms of action. Further, patients will be subjected to oral and rectal swabs, and urine sampling to determine virus shedding. The patients will be monitored for time to progression, progression free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Have histologic or cytologic evidence of colorectal carcinoma (CRC), pancreatic carcinoma (PC), biliary cancer, or epithelial ovarian carcinoma (EOC which may encompass epithelial ovarian, fallopian tube or primary peritoneal carcinoma).
2. Have advanced disease, defined as cancer that is either metastatic or locally advanced, unresectable, and for which radiotherapy or other locoregional therapies are not considered treatment of choice but systemic chemotherapy or no therapy is planned.
3. Have one of the following treatment situations apply:

   1. Colorectal carcinoma (CRC) I. A patient with refractory or recurrent metastatic CRC who has either received all conventional therapy; or is entering a "resting" phase between reasonable conventional treatments. II. A patient who is amenable to treatment with LOAd703 plus gemcitabine as a single agent conditioning regimen.
   2. Pancreatic cancer I. A patient with either locally advanced, unresectable or metastatic disease who is eligible to receive any line of conventional treatment consisting of gemcitabine and/or nab-paclitaxel. II. A patient who is amenable to treatment with LOAd703 as an "add-on" to standard-of-care gemcitabine-based or nab-paclitaxel- based regimens or gemcitabine or nab-paclitaxel as single agents. c. Biliary cancer I. A patient with either locally advanced unresectable or metastatic biliary cancer who is either treatment-naïve or has received any number of lines of treatment. II. Patient who is amenable to treatment with LOAd703 as an "add-on" to standard-of-care treatment consisting of gemcitabine combined with other agents (e.g. gemcitabine/low-dose cisplatin, gemcitabine/oxaliplatin, etc) in the first line setting or gemcitabine in a combination regimen or as a single agent in latter lines of treatment. d. Ovarian Cancer I. A patient with either epithelial ovarian, fallopian tube or primary peritoneal carcinoma.

   II. The patient has either:

   i) Residual disease following first-line standard-of-care combination chemotherapy. ii) Platinum-sensitive disease (platinum free interval ≥ 6 months) in early relapse following first-line standard-of care combination chemotherapy. iii) Platinum-resistant disease and received at least 3 lines of standard treatment. These treatments should have included bevacizumab and/or PARP inhibitors if they are reasonable candidates for such. III. Amenable to treatment with LOAd703 as an "add-on" to standard-of-care paclitaxel-based regimens (excluding bevacizumab), paclitaxel as a single agent, or gemcitabine as a single agent.
4. Have a disease burden that is considered low (i.e. low tumor burden), which is defined on a patient-by-patient basis as per principal investigator's discretion. A rough guideline for defining low tumor burden is that the sum of the product of the bidimensional measurements for all lesions is < 70 cm2.
5. Have a measurable disease by standard imaging techniques per RECIST criteria. Measurable lesions must be outside of any prior radiation field(s), unless disease progression has been documented at that disease site subsequent to radiation.
6. At least one non-irradiated (or irradiated but disease progression documented at the site subsequent to radiation) lesion must be suitable for image-guided intratumoral injection and needle biopsy.
7. Be medically suited to sedation if required during intratumoral injections.
8. Be at least 18 years-old.
9. Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2.
10. Have no remaining acute toxic effects from previous anticancer therapy > grade 1 except for any grade of alopecia.
11. Have adequate baseline organ/hematological function, as demonstrated by the following:

    1. Absolute neutrophil count (ANC) ≥1.0 x 109/l
    2. Hemoglobin ≥9 g/dl
    3. Platelet count ≥ 100 x 109/l
    4. Bilirubin < 1.5 times the institutional upper limit of normal (ULN)
    5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <2.5 (3, if liver metastases are present) times the institutional ULN.
    6. Serum creatinine <2 times the institutional ULN or calculated creatinine clearance >35 mL/min
    7. Prothrombin (INR)<1.5 or prothrombin time (PT) <1.5 ULN; and either partial thromboplastin time or activated partial thromboplastin time (PTT or aPTT) ≤ 1.5 times the ULN.
12. The patient must understand and be willing to provide written informed consent.

Exclusion Criteria:

1. Any concurrent treatment that would compromise the study including but not limited to continuous high dose corticosteroids (>0.5mg/kg), lymphodepleting antibodies or cytotoxic agents.
2. Treatment with high dose immune inhibitors including lymphotoxic monoclonal antibodies such as alemtuzumab (CampathR), or sirolimus (RapamuneR) and its analogs, biological therapy, cytotoxic agents or any investigational agents within 21 days of registration.
3. Ovarian carcinoma patients should not be eligible to PARP inhibitor treatment.
4. Patients on warfarin (or other anti-coagulants) are not eligible.
5. Women who are pregnant, lactating, or planning to become pregnant during the study period, or women of childbearing potential who are not using acceptable contraceptive methods. A woman is considered of childbearing potential if she is not surgically sterile or is less than 1 year since last menstrual period. Acceptable contraceptive methods are: combined (estrogen and progesterone containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progesterone-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion and vasectomized partner.
6. Men who do not consent to the use of condom during intercourse during study participation.
7. Known active hepatitis B or C infection, or HIV infection.
8. Patients with active, severe, autoimmune disease.
9. Uncontrolled intercurrent illness including but not limited to psychiatric illness/social situations that in the opinion of the Investigator would compromise compliance of study requirements or put the patient at unacceptable risk.
10. Other malignancies within the past 2 years (not including basal and squamous cell carcinoma of the skin, localized prostate cancer or in situ cervix carcinoma).
11. Patients must agree to not to vaccinate with living vaccines during participation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2023-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angelica Loskog, PhD, Study Chair — Lokon Pharma AB
Locations (2):
- Sweden (2):
  - Karolinska University Hospital, Huddinge, Stockholm
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Overall, a total of 47 subjects signed the informed consent, 5 out of 47 subjects were screening failures and 42 subjects were assigned to the study treatment (Group 1, 2 or 3). One subject was assigned to Group 3, but was not exposed to the study treatment.
Groups:
- Group 1 LOAd703 5x10e10 VP + SOC Tailored to the Indication: LOAd703 (5x10e10 VP) oncolytic adenovirus administered add-on to standard of care chemotherapy or gemcitabine immune-conditioning if standard of care is no longer an option (e.g. after last line)
  LOAd703: Oncolytic adenovirus serotype 5/35 encoding TMZ-CD40L and 4-1BBL
- Group 2 LOAd703 1x10e11 VP + SOC Tailored to the Indication: LOAd703 (1x10e11 VP) oncolytic adenovirus administered add-on to standard of care chemotherapy or gemcitabine immune-conditioning if standard of care is no longer an option (e.g. after last line)
  LOAd703: Oncolytic adenovirus serotype 5/35 encoding TMZ-CD40L and 4-1BBL
- Group 3 LOAd703 5x10e11 VP + SOC Tailored to the Indication: LOAd703 (5x10e11 VP) oncolytic adenovirus administered add-on to standard of care chemotherapy or gemcitabine immune-conditioning if standard of care is no longer an option (e.g. after last line)
  LOAd703: Oncolytic adenovirus serotype 5/35 encoding TMZ-CD40L and 4-1BBL
Period: Group 1: LOAd703 Dose Level 5x10e10VP
Arm/Group | Group 1 LOAd703 5x10e10 VP + SOC Tailored to the Indication | Group 2 LOAd703 1x10e11 VP + SOC Tailored to the Indication | Group 3 LOAd703 5x10e11 VP + SOC Tailored to the Indication
Started | 3 | 0 | 0
Completed | 1 | 0 | 0
Not Completed | 2 | 0 | 0
Not completed — Progressive Disease | 2 | 0 | 0
Period: Group 2: LOAd703 Dose Level 1x10e11 VP
Arm/Group | Group 1 LOAd703 5x10e10 VP + SOC Tailored to the Indication | Group 2 LOAd703 1x10e11 VP + SOC Tailored to the Indication | Group 3 LOAd703 5x10e11 VP + SOC Tailored to the Indication
Started | 0 | 12 | 0
Completed | 0 | 2 | 0
Not Completed | 0 | 10 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Progressive Disease | 0 | 7 | 0
Not completed — Other Reason | 0 | 1 | 0
Period: Group 3: LOAd703 Dose Level 5x10e11VP
Arm/Group | Group 1 LOAd703 5x10e10 VP + SOC Tailored to the Indication | Group 2 LOAd703 1x10e11 VP + SOC Tailored to the Indication | Group 3 LOAd703 5x10e11 VP + SOC Tailored to the Indication
Started | 0 | 0 | 27
Completed | 0 | 0 | 1
Not Completed | 0 | 0 | 26
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Death | 0 | 0 | 4
Not completed — Progressive Disease | 0 | 0 | 16
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Not Exposed to LOAd703 | 0 | 0 | 1
Not completed — Other Reason | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 LOAd703 5x10e10 VP + SOC Tailored to the Indication | Group 2 LOAd703 1x10e11 VP + SOC Tailored to the Indication | Group 3 LOAd703 5x10e11 VP + SOC Tailored to the Indication | Total
Number analyzed (Participants) | 3 | 12 | 27 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (12.7) | 62.9 (12.4) | 63.1 (8.1) | 62.5 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 6 | 17 | 23
  Male | 3 | 6 | 10 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 12 | 27 | 42
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 3 | 12 | 27 | 42
ECOG score [Number; unit: participants] — ECOG 0= Fully active, able to carry on all pre-disease performance without restriction; ECOG 1= Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; ECOG 2= Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours; ECOG 3= Capable of only limited self-care, confined to bed or chair more than 50% of waking hours; ECOG 4= Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair; ECOG 5= Dead.
  participants
    ECOG score 0 | 1 | 4 | 21 | 26
    ECOG score 1 | 2 | 7 | 6 | 15
    ECOG score 2 | 0 | 1 | 0 | 1
Cancer Diagnosis [Number; unit: participants]
  Pancreatic cancer | 1 | 9 | 19 | 29
  Colorectal carcinoma | 2 | 2 | 1 | 5
  Ovarian cancer | 0 | 1 | 4 | 5
  Biliary cancer | 0 | 0 | 3 | 3
Current oncological disease [Number; unit: participants] — Locally advanced (cancer that has spread from where it started to nearby tissue or lymph nodes); metastatic (spread of cancer from the primary site to other places in the body)
  participants
    Locally advanced | 0 | 4 | 4 | 8
    Metastatic | 3 | 8 | 23 | 34

OUTCOME MEASURES:

1. Primary Outcome: Safety: Toxicity Symptoms Graded According to CTCAE v4.03.
Description: The toxicity symptoms were graded according to CTCAE v4.03.
Time Frame: Up to 50 weeks
Population: Overall, a total of 42 subjects were assigned to the study treatment, 1 out of 42 did not receive the study treatment and it was not included in the safety evaluation. The subject who did not receive the study treatment was assigned to group 3.
Measure: Number; unit: Number of Events
Arm/Group | Group 1 LOAd703 5x10e10 VP + SOC Tailored to the Indication | Group 2 LOAd703 1x10e11 VP + SOC Tailored to the Indication | Group 3 LOAd703 5x10e11 VP + SOC Tailored to the Indication
Number analyzed (Participants) | 3 | 12 | 26
Number of Events
  All adverse events (AE) | 61 | 139 | 411
  All serious adverse events (SAEs) | 7 | 31 | 63
  Serious adverse reactions (SARs) related to LOAd703 | 3 | 4 | 21
  AE leading to withdrawal from the study | 0 | 1 | 2
  AE leading to LOAd703 discontinuation | 0 | 2 | 6
  AE leading to death | 0 | 0 | 1
  AE related to LOAd703 | 29 | 33 | 169
  AE related to LOAd703 grade 1 | 15 | 29 | 111
  AE related to LOAd703 grade 2 | 14 | 3 | 52
  AE related to LOAd703 grade 3 | 0 | 0 | 6
  AE related to LOAd703 grade 4 | 0 | 1 | 0
  AE related to LOAd703 grade 5 | 0 | 0 | 0
  AE unrelated to LOAd703 | 32 | 106 | 242

2. Primary Outcome: Immune Reactions to LOAd703 Virus as Assessed by Anti-adenovirus Ig ELISA
Description: Fold change between baseline and evaluation visit for anti-adenovirus antibodies (LOAd703).
  The baseline is the last available measurement taken before the first LOAd703 treatment. Evaluation is a measurement taken from subjects receiving at least 3 LOAd703 treatments.
Time Frame: Up to 50 weeks
Measure: Mean (Standard Deviation); unit: fold change
Groups:
- LOAd703 Dose 5x10e10 VP: LOAd703 (5x10e10 VP) oncolytic adenovirus administered add-on to standard of care chemotherapy or gemcitabine immune-conditioning if standard of care is no longer an option (e.g. after last line)
  LOAd703: Oncolytic adenovirus serotype 5/35 encoding TMZ-CD40L and 4-1BBL
- LOAd703 Dose 1x10e11 VP: LOAd703 (1x10e11 VP) oncolytic adenovirus administered add-on to standard of care chemotherapy or gemcitabine immune-conditioning if standard of care is no longer an option (e.g. after last line)
  LOAd703: Oncolytic adenovirus serotype 5/35 encoding TMZ-CD40L and 4-1BBL
- LOAd703 Dose 5x10e11 VP: LOAd703 (5x10e11 VP) oncolytic adenovirus administered add-on to standard of care chemotherapy or gemcitabine immune-conditioning if standard of care is no longer an option (e.g. after last line)
  LOAd703: Oncolytic adenovirus serotype 5/35 encoding TMZ-CD40L and 4-1BBL
Arm/Group | LOAd703 Dose 5x10e10 VP | LOAd703 Dose 1x10e11 VP | LOAd703 Dose 5x10e11 VP
Number analyzed (Participants) | 3 | 12 | 24
fold change | 41.63 (8.39) | 15.81 (10.33) | 31.77 (24.31)

3. Secondary Outcome: Response on Tumor Size by Dose and Cancer Diagnosis
Description: Local and distant anti-tumoral size changes assessed by appropriate imaging accordingly to RECIST 1.1. Complete Response (CR), complete macroscopic disappearance of all tumors; Partial Response (PR), a reduction of at least 30% in the sum of all tumor diameters from baseline; one/more lesions fulfilling the criteria for PR and other/others for progressive disease (PD); Stable disease (SD), Neither PR nor PD; Progressive disease (PD), at least 20% increase in the sum of all tumor diameters from the smallest tumor size and/or the appearance of new tumor lesion/s; Overall response rate (ORR) = CR + PR; Clinical benefit rate (CBR) = CR + PR + SD.
Time Frame: Up to 50 weeks
Population: Response on tumor size was evaluated in participants who have received at least 3 doses of LOAd703 and performed computed tomography (CT) evaluation at baseline and at week 9 (Visit 5). Group 1 (5x10e10 VP): all the 3 participants met the criteria to be included in this analysis; Group 2 (1x10e11 VP): from a total of 12 participants, 10 met the criteria to be included in this analysis; Group 3 (5x10e11 VP): from a total of 27 participants, 22 met the criteria to be included in this analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Colorectal Cancer: Response on tumor size by cancer diagnosis for colorectal cancer.
- Biliary Cancer: Response on tumor size by cancer diagnosis for biliary cancer.
- Pancreatic Cancer: Response on tumor size by cancer diagnosis for pancreatic cancer.
- Ovarian Cancer: Response on tumor size by cancer diagnosis for ovarian cancer.
Arm/Group | LOAd703 Dose 5x10e10 VP | LOAd703 Dose 1x10e11 VP | LOAd703 Dose 5x10e11 VP | Colorectal Cancer | Biliary Cancer | Pancreatic Cancer | Ovarian Cancer
Number analyzed (Participants) | 3 | 10 | 22 | 5 | 3 | 24 | 3
Participants
  Complete response (CR) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial response (PR) | 0 | 3 | 3 | 0 | 0 | 6 | 0
  Stable disease (SD) | 1 | 4 | 11 | 2 | 1 | 11 | 2
  Progressive disease (PD) | 2 | 3 | 8 | 3 | 2 | 7 | 1
  Overall response rate (ORR) | 0 | 3 | 3 | 0 | 0 | 6 | 0
  Clinical benefit rate (CBR) | 1 | 7 | 14 | 2 | 1 | 17 | 2

4. Secondary Outcome: Overall Survival
Description: Months of overall survival (OS) from registration by dose and cancer diagnosis
Time Frame: From registration date to date of death, assessed up to 40 months
Population: OS was evaluated in participants who have received at least 3 doses of LOAd703 and performed computed tomography (CT) evaluation at baseline and at week 9 (Visit 5). Group 1 (5x10e10 VP): all the 3 participants met the criteria to be included in this analysis; Group 2 (1x10e11 VP): from a total of 12 participants, 10 met the criteria to be included in this analysis; Group 3 (5x10e11 VP): from a total of 27 participants, 22 met the criteria to be included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LOAd703 Dose 5x10e10 VP | LOAd703 Dose 1x10e11 VP | LOAd703 Dose 5x10e11 VP | Colorectal Cancer | Biliary Cancer | Pancreatic Cancer | Ovarian Cancer
Number analyzed (Participants) | 3 | 10 | 22 | 5 | 3 | 24 | 3
Months | 4.40 [3.02 to 12.85] | 8.44 [2.66 to 40.54] | 7.38 [5.39 to 10.71] | 5.36 [3.02 to 8.44] | 6.64 [5.26 to 7.46] | 7.29 [5.39 to 12.85] | 40.54 [9.69 to 40.54]

5. Secondary Outcome: Time to Progression
Description: Time to progression from registration by dose and cancer diagnosis
Time Frame: From registration date to date of progression, assessed up to 40 months
Population: Time to progression was evaluated in participants who have received at least 3 doses of LOAd703 and performed computed tomography (CT) evaluation at baseline and at week 9 (Visit 5). Group 1 (5x10e10 VP): all the 3 participants met the criteria to be included in this analysis; Group 2 (1x10e11 VP): from a total of 12 participants, 10 met the criteria to be included in this analysis; Group 3 (5x10e11 VP): from a total of 27 participants, 22 met the criteria to be included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LOAd703 Dose 5x10e10 VP | LOAd703 Dose 1x10e11 VP | LOAd703 Dose 5x10e11 VP | Colorectal Cancer | Biliary Cancer | Pancreatic Cancer | Ovarian Cancer
Number analyzed (Participants) | 3 | 10 | 22 | 5 | 3 | 24 | 3
Months | 2.40 [1.74 to 3.68] | 3.79 [1.81 to 5.49] | 3.88 [1.87 to 5.72] | 2.40 [1.74 to 3.84] | 1.81 [1.58 to 4.76] | 3.75 [2.27 to 5.72] | 3.88 [1.87 to 20.07]

6. Secondary Outcome: Progression Free Survival
Description: Months of progression free survival (PFS) from registration by dose and cancer diagnosis
Time Frame: From registration date to date of progression, or date of death, which ever came first, assessed up to 40 months
Population: PFS was evaluated in participants who have received at least 3 doses of LOAd703 and performed computed tomography (CT) evaluation at baseline and at week 9 (Visit 5). Group 1 (5x10e10 VP): all the 3 participants met the criteria to be included in this analysis; Group 2 (1x10e11 VP): from a total of 12 participants, 10 met the criteria to be included in this analysis; Group 3 (5x10e11 VP): from a total of 27 participants, 22 met the criteria to be included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LOAd703 Dose 5x10e10 VP | LOAd703 Dose 1x10e11 VP | LOAd703 Dose 5x10e11 VP | Colorectal Cancer | Biliary Cancer | Pancreatic Cancer | Ovarian Cancer
Number analyzed (Participants) | 3 | 10 | 22 | 5 | 3 | 24 | 3
Months | 2.40 [1.74 to 3.68] | 3.79 [1.81 to 5.49] | 4.32 [1.87 to 5.72] | 2.40 [1.74 to 5.36] | 1.81 [1.58 to 4.76] | 4.62 [2.27 to 5.72] | 3.88 [1.87 to 20.07]

7. Secondary Outcome: Systemic Immune Activation
Description: Percentage of participants with upregulated immune marker in blood at evaluation as compared to baseline.
  The baseline is the last available measurement taken before the first LOAd703 treatment. Evaluation is a measurement taken from subjects receiving at least 3 LOAd703 treatments.
Time Frame: Up to 50 weeks
Measure: Number; unit: Percentage of Participants
Arm/Group | LOAd703 Dose 5x10e10 VP | LOAd703 Dose 1x10e11 VP | LOAd703 Dose 5x10e11 VP
Number analyzed (Participants) | 3 | 11 | 25
Percentage of Participants | 100 | 100 | 100

8. Secondary Outcome: Immune Cell Activation
Description: Fold change between baseline and evaluation visit for CD8+ CD3+ T cells activation evaluated by flow cytometry.
  The baseline is the last available measurement taken before the first LOAd703 treatment. Evaluation is a measurement taken from subjects receiving at least 3 LOAd703 treatments.
Time Frame: Up to 50 weeks
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | LOAd703 Dose 5x10e10 VP | LOAd703 Dose 1x10e11 VP | LOAd703 Dose 5x10e11 VP
Number analyzed (Participants) | 3 | 11 | 25
fold change | 1.01 (0.39) | 1.19 (0.32) | 1.17 (0.48)

9. Secondary Outcome: Presence of LOAd703 Virus in Blood
Description: Percentage of PK samples analyzed that were positive for viral DNA/ml in serum.
Time Frame: Up to 50 weeks
Measure: Number; unit: Percentage of positive samples
Units Other Than Participants: Blood samples
Arm/Group | LOAd703 Dose 5x10e10 VP | LOAd703 Dose 1x10e11 VP | LOAd703 Dose 5x10e11 VP
Number analyzed (Participants) | 3 | 12 | 26
Number analyzed (Blood samples) | 18 | 93 | 186
Percentage of positive samples | 22.22 | 16.13 | 35.48

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the first LOAd703/chemotherapy treatment up to 50 weeks (final follow-up). All-Cause Mortality was assessed from registration date to date of death, assessed up to 40 months.
Description: The number of participants with adverse events and not the number of events are reported.
Arm/Group | Group 1 LOAd703 5x10e10 VP + SOC Tailored to the Indication | Group 2 LOAd703 1x10e11 VP + SOC Tailored to the Indication | Group 3 LOAd703 5x10e11 VP + SOC Tailored to the Indication
All-Cause Mortality (participants affected / at risk) | 3/3 | 10/12 | 23/26
Serious Adverse Events (participants affected / at risk) | 3/3 | 12/12 | 20/26
Other Adverse Events (participants affected / at risk) | 3/3 | 11/12 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 LOAd703 5x10e10 VP + SOC Tailored to the Indication (N=3) | Group 2 LOAd703 1x10e11 VP + SOC Tailored to the Indication (N=12) | Group 3 LOAd703 5x10e11 VP + SOC Tailored to the Indication (N=26)
Pyrexia (General disorders) | 1 | 1 | 11
Fatigue (General disorders) | 1 | 0 | 1
General physical health deterioration (General disorders) | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 2 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 2
Cytokine release syndrome (Immune system disorders) | 0 | 1 | 4
Clostridial infection (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 2 | 1
Liver abscess (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 4
Pneumonia (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 1
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1
Device dislocation (Product Issues) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1
Glomerulonephritis membranoproliferative (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 LOAd703 5x10e10 VP + SOC Tailored to the Indication (N=3) | Group 2 LOAd703 1x10e11 VP + SOC Tailored to the Indication (N=12) | Group 3 LOAd703 5x10e11 VP + SOC Tailored to the Indication (N=26)
Anaemia (Blood and lymphatic system disorders) | 1 | 4 | 8
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 3 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 2 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Periorbital oedema (Eye disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 4
Nausea (Gastrointestinal disorders) | 2 | 5 | 16
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 10
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 5
Ascites (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 6
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2
Change of bowel habit (Gastrointestinal disorders) | 0 | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 2
Gingival blister (Gastrointestinal disorders) | 0 | 0 | 1
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 0 | 1
Chills (General disorders) | 3 | 3 | 11
Fatigue (General disorders) | 2 | 7 | 16
General physical health deterioration (General disorders) | 1 | 0 | 2
Malaise (General disorders) | 1 | 0 | 1
Oedema peripheral (General disorders) | 2 | 5 | 6
Pyrexia (General disorders) | 3 | 8 | 24
Discomfort (General disorders) | 0 | 1 | 0
Gastroenteritis (General disorders) | 0 | 1 | 0
Injection site oedema (General disorders) | 0 | 1 | 0
Localised oedema (General disorders) | 0 | 1 | 1
Face oedema (General disorders) | 0 | 0 | 1
Feeling cold (General disorders) | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 1
Injection site inflammation (General disorders) | 0 | 0 | 1
Injection site pain (General disorders) | 0 | 0 | 2
Mucosal inflammation (General disorders) | 0 | 0 | 2
Pain (General disorders) | 0 | 0 | 1
Swelling (General disorders) | 0 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 2
Clostridial infection (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 1
Infection (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2 | 2
Oral candidiasis (Infections and infestations) | 0 | 1 | 0
Oral fungal infection (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 1
Groin infection (Infections and infestations) | 0 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Peripancreatic fluid collection (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 4
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 2
C-reactive protein increased (Investigations) | 0 | 2 | 6
Cardiac murmur (Investigations) | 0 | 1 | 0
Electrocardiogram abnormal (Investigations) | 0 | 1 | 0
Heart rate irregular (Investigations) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 2
Neutrophil count decreased (Investigations) | 0 | 1 | 5
Weight decreased (Investigations) | 0 | 1 | 3
White blood cell count decreased (Investigations) | 0 | 1 | 5
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 3
Blood albumin decreased (Investigations) | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 2
Blood pressure decreased (Investigations) | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Tumour thrombosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 2 | 6
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 2
Urinary tract infection (Renal and urinary disorders) | 0 | 3 | 3
Glomerulonephritis membranoproliferative (Renal and urinary disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Hypertension (Vascular disorders) | 2 | 2 | 4
Hypotension (Vascular disorders) | 0 | 2 | 3
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 2
Embolism (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-12-21): https://cdn.clinicaltrials.gov/large-docs/89/NCT03225989/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/89/NCT03225989/SAP_001.pdf